CLINICAL TRIAL: NCT06789016
Title: Dexmedetomidine for ESPB in Pain Management After Pediatric Idiopathic
Brief Title: Dexmedetomidine for ESPB in Pain Management After Pediatric Idiopathic Scoliosis Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/2024
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-09

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXMEDETOIDINE (Active Comparator): 0.2% ropivacaine 0.5ml/kg+ 0.1ug/kg Dexamethasone for erector spinae plane block
  Interventions: Drug: Dexmedetomidine
- CONTROL (Active Comparator): 0.2% ropivacaine 0.5ml/kg for erector spinae plane block
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: Dexmedetomidine — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1ug/kg Dexmedetomidine for the erector spine plane block
  Other Names: DEX
  Arms: DEXMEDETOIDINE
Drug: 0.9%NaCl — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the erector spine plane block
  Other Names: saline
  Arms: CONTROL

SUMMARY:
Effect of perineurial dexmedetomidine on erector spinal plane block duration for pediatric, idiopathic scoliosis surgery.

DETAILED DESCRIPTION:
This study proposes to explore the effect of perineurial Dexmedetomidine on the duration of erector spinal plane block for pediatric idiopathic scoliosis surgery.

Children need good analgesia after scoliosis surgery. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexmedetomidine, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for idiopathic scoliosis surgery
* age >10 and <18 years

Exclusion Criteria:

* age < 10 years
* age < 18 years
* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
First need of opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours after surgery
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Nerve damage [range 0-4] | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
adverce effects | durring surgery
  nausea, vomitting, bradycardia, hypotension
adverce effects | 48 hours after surgery
  nausea, vomitting, bradycardia, hypotension
MEP | durring surgery
  motor evoced potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes